CLINICAL TRIAL: NCT03696979
Title: The Effect of Myofascial Induction and Therapeutic Pain Education in Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Mehmet ÜNAL, director physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 76678999
Record Dates: First submitted 2018-09-21; First posted 2018-10-05 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Back Pain
MeSH Terms: conditions — Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- myofascial induction (Active Comparator): Twice a week for 8 weeks. Lumbar interfacial field stroke application, Lumbar interfacial field to deep application, Lumbar region cross-hands induction technique, Hip flexor region induction.
  Interventions: Other: Myofascial induction therapy
- Therapeutic Pain education (Active Comparator): Pain education,twice a week for 8 weeks. The mechanism of pain,Pain processing in the center, How sensitive the central nervous system is in chronic pain, Pain becomes chronic with the contribution of factors, Problems related to fear of pain will be explained in detail.
  Interventions: Other: Therapeutic pain education

INTERVENTIONS:
Other: Myofascial induction therapy — Myofascial induction therapy is a therapy concept focused on optimizing function and balance within the fascial system. The approach aims at global recovery, local correction and painless body use.
  Arms: myofascial induction
Other: Therapeutic pain education — Therapeutic pain education is a training intervention that aims to reduce pain and disability by helping patients better understand the biological processes that support pain states. The neurobiology of pain and pain processed by the nervous system is explained to the patient in detail. Changes the patient's olab viewpoint to pain. For example, the patient believes that the cause of pain is caused by tissue damage. The patient who receives pain training understands that the cause of pain is the hypersensitive central nervous system. As a result, the patient's fear avoidance behavior decreases and he starts to move more easily. Because the sensitivity of the central nervous system will be alleviated, the perceived pain will decrease.
  Arms: Therapeutic Pain education

SUMMARY:
The aim of this study was to investigate the effects of therapeutic pain education and myofascial induction therapy on pain and function in patients with chronic low back pain. In the literature, studies on myofascial induction therapy in patients with chronic low back pain are very limited and there is no study comparing therapeutic pain training.

DETAILED DESCRIPTION:
Lumbar pain has become a major health problem which is growing and is very common in all societies and negatively affects the full well-being of the individual. It has been reported that 80% of the population experienced low back pain at any time in their lives. The prolongation of this painful process affects the physical, mental and psychological state of the patient and limits its daily functions. The acute or chronic pain determines the nature and duration of pain. Low back pain lasting 12 weeks or more is defined as chronic. In chronic diseases, lumbar pain, which is the first one, restricts the daily activities of the person due to current chronic pain or deterioration of functional status and causes loss of labor force.

Myofascial induction therapy is a therapy concept focused on optimizing function and balance within the fascial system. The approach aims at global recovery, local correction and painless body use.

Superficial procedures are directed to surface and / or local restrictions that can be directly detected by palpation. Deep myofascial induction therapy is a method that eliminates the limitations of the myofascial system and the three-dimensional pressures.

Therapeutic pain education is a training intervention that aims to reduce pain and disability by helping patients better understand the biological processes that support pain states. The neurobiology of pain and pain processed by the nervous system is explained to the patient in detail. Changes the patient's olab viewpoint to pain. For example, the patient believes that the cause of pain is caused by tissue damage. The patient who receives pain education understands that the cause of pain is the hypersensitive central nervous system. As a result, the patient's fear avoidance behavior decreases and he starts to move more easily. Because the sensitivity of the central nervous system will be alleviated, the perceived pain will decrease.

ELIGIBILITY:
Inclusion Criteria:

* Between 25-65 years old
* Low back pain for at least 12 weeks
* Physical therapy in the last 1 month
* There is no other disease that may cause low back pain.

Exclusion Criteria:

* Stem pressure associated with pain
* Having severe discopathy
* Available compression fracture
* To have rheumatic or inflammatory disease that may cause back pain.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-11-20 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2020-02-10 (Actual)

PRIMARY OUTCOMES:
Mc Gill pain survey | 8 week
  The McGill Pain Questionnaire (MPQ) is a self-reporting measure of pain used for patients with a number of diagnoses. It assesses both quality and intensity of subjective pain. Seven words are selected from the following categories: dimension 1 to 10 (pain descriptors), three words; dimensions 11 to 15 (affective components of pain), dimension 16 (evaluation of pain) one word, and dimension 17 to 20 (miscellaneous) one word. Scores are tabulated by summing values associated with each word; scores range from 0 (no pain) to 78 (severe pain). Qualitative differences in pain may be reflected in respondent's word choice
Roland Morris Disability index | 8 week
  Roland-Morris Disability Questionnaire[1] is designed to assess self-rated physical disability caused by low back pain. There are different questionnaires available, which differ from each other in the number of statements: 24-, 18- and 11-item questionnaire. The patient is asked to tick a statement when it applies to him that specific day, this makes it possible to follow changes in time. The end score is the sum of the ticked boxes. The score ranges from 0 (no disability) to 11, 18 or 24 (max. disability) depending on the questionnaire that is used.
Survey of fear avoidance beliefs | 8 week
  The Fear-Avoidance Beliefs Questionnaire (FABQ) is a patient reported questionnaire which specifically focuses on how a patient's fear avoidance beliefs about physical activity and work may affect and contribute to their low back pain and resulting disability. The questionnaire consists of 16 items in which a patient rates their agreement with each statement on a 7-point Likert scale. Where 0= completely disagree, 6=completely agree. There is a maximum score of 96.
Evaluation of mobility (finger ground test) | 8 week
  fingertip-to-floor (FTF) test as an outcome measure on the great majority of my patients presenting with lumbo-pelvic pain, for the simple reason that forward bending is one of the more painful and limited movements, especially in those with neural symptoms.
  The FTF test has been shown to have excellent reliability without the use of standardized instructions and patient positioning.
  It must be stated that the FTF test has been criticized for not measuring isolated lumbar flexion range of motion, with the argument that forward bending range is also based on pelvic, hip, thoracic spine, dural and shoulder mobility.
SF.36 Healthy life survey | 8 week
  The Short Form (36) Health Survey is a multi-purpose survey designed to capture adult patients' perceptions of their own health and well-being. Based on a much longer survey developed in the 1980's by Ware, J.E., the SF-36 has 36 items grouped in 8 dimensions: physical functoning, physicial and emotional limitations, social functioning, bodily pain, general and mental health.
Ultrasound examination of thoracolumbar fascia | 8 week
  thoracolumbar fascia Measurements and evaluation of TLF were obtained using single blind method when investigator didn't know any clinical information about a patient. Thickness of TLF was measured from both sides of a spine in the direction perpendicular to the skin. According to methodic of Langevin mentioned above TLF was divided to subdermal (SD) and supramuscular (SM). The general thickness of TLF is defined as the distance between deep border of the dermis and the superficial border of the muscle. TLF is hyperechogenic one or several layers (planes) structure which thickness is measured as a distance between the muscle and subdermal part of fascia.

CONTACTS AND LOCATIONS:
Locations (1):
- Mehmet Unal, Kocaeli, Select..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided